CLINICAL TRIAL: NCT07162246
Title: Combined Gamma Knife/Linac Hypofractionated Stereotactic Radiosurgery for Large Intracranial VolumEs (GK-LIVE): A Prospective Phase II Single-Arm Trial
Brief Title: Combined Gamma Knife/Linac Radiosurgery for Large Brain Tumors / Metastases
Acronym: GK-LIVE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GK-LIVE
Record Dates: First submitted 2025-08-07; First posted 2025-09-09 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-08

CONDITIONS: Brain (Nervous System) Cancers; Brain Metastasases; SRS
MeSH Terms: conditions — Neurologic Manifestations; Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Arm (Experimental)
  Interventions: Radiation: Radiation Therapy

INTERVENTIONS:
Radiation: Radiation Therapy — Adaptive radiation therapy with GK boost

SUMMARY:
When cancer spreads to the brain, doctors often use a precise type of radiation therapy called stereotactic radiosurgery (SRS) to treat these tumors. This treatment can effectively control brain tumors while helping protect healthy brain tissue. However, when brain tumors or the areas where tumors were surgically removed are larger, treatment outcomes in terms of side effects and tumour control can become worse. Specifically, standard SRS on larger areas can have lower tumour control and higher risk of side effects, particularly a condition called radiation necrosis, which can cause swelling and damage in nearby healthy brain tissue.

Currently at Sunnybrook, large brain tumors are typically treated with SRS spread over 5 daily treatments using a machine called a linear accelerator. While this approach works well for many patients, it may be possible to improve results by combining two different types of radiation therapy machines - the linear accelerator and another specialized machine called the Gamma Knife.

In this study, the investigators want to test a new treatment approach where patients first receive 4 daily treatments using the linear accelerator, followed by a 1-2 week break, and then a final treatment using the Gamma Knife. The break between treatments allows the study doctors to take new scans and precisely target any remaining tumor, which may shrink during the break, thereby potentially reducing the amount of healthy brain tissue exposed to radiation. The Gamma Knife is also particularly good at delivering very precise radiation while sparing nearby healthy tissue. Lastly, there may be unique biological mechanisms between the two technologies that could be taken advantage of, by combining the technologies in the participant's treatment plan, to improve cancer control.

The investigators believe this combined approach might help achieve better tumor control while reducing the risk of side effects compared to using just the linear accelerator. This study will help the investigators understand if this new treatment strategy is safe and effective for patients with large brain tumors or surgical cavities, and whether it leads to better outcomes than the current treatment approach.

ELIGIBILITY:
Inclusion Criteria:

* Presence of up to two large intracranial lesions
* Up to 10 (previously untreated, or progressing after previous treatment) brain metastases at the time of enrollment on the diagnostic MRI (which includes the ILLs) to be treated with SRS/HSRS
* Age => 18 years
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Expected survival >3 months
* Patients that are deemed suitable for both GK and Linac based treatment
* Patients that are able to hold systemic cancer chemotherapy/immunotherapy at least 2 days prior and following an SRS fraction

Exclusion Criteria:

* Prior SRS to the ILLs
* Prior WBRT, or plan for concurrent WBRT with the protocol treatment
* Presence or history of any leptomeningeal/pachymeningeal disease
* Metastatic disease within the ventricles of the brain or corpus callosum
* Small cell, hematopoietic or germ cell primaries
* Patient with absolutely contraindications for MRI
* Severe symptoms that preclude MRI or treatment using standard procedures for Linac or GK
* Pregnant or lactating patient
* Inability or unwillingness to undergo informed consent or post-treatment follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-07-14 (Actual); Primary Completion 2029-06 (Estimated); Study Completion 2030-06 (Estimated)

PRIMARY OUTCOMES:
Cumulative incidence of late local complication (LLC) | From end of protocol treatment to development of local failure or symptomatic ISRS Grade => 2 radionecrosis (assessed up to 24 months)

SECONDARY OUTCOMES:
Overall Survival | Completion of protocol treatment to date of death (assessed up to 24 months)
Distant Brain Progression-Free Survival | Date of protocol treatment to either appearance of additional metastatic disease within the brain, or death (assessed up to 24 months)
Cumulative Incidence of Local Failure | Date of completion of protocol treatment to local failure (assessed up to 24 months)
Cumulative Incidence of Radiation Necrosis | Date of protocol treatment to development of symptomatic radiation necrosis (assessed up to 24 months)
Treatment-Related Toxicity | Throughout study participation and assessed up to 24 months following treatment completion
  From changes to baseline, as defined by CTCAE v5.0
Change in Neurological Function | From enrollment onwards, up until 24 months after protocol treatment completion
  Through changes in the NANO scale
Health-Related Quality of Life | From enrollment onwards, up until 24 months after protocol treatment completion
  Through changes in responses to health-related quality of life surveys completed during study participation

CONTACTS AND LOCATIONS:
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided